CLINICAL TRIAL: NCT06308900
Title: Evaluation of Non-technical Skills of Clinical Simulation in Physiotherapy Students and Analysis of the Experience
Brief Title: Non-technical Skills of Clinical Simulation in Physiotherapy Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Hernández-Guillén, Principal investigator, University of Valencia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CL_SIMULATION_01
Record Dates: First submitted 2024-03-05; First posted 2024-03-13 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Healthy
Keywords: Physiotherapy; Students; Learning methodology; Clinical simulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Physitherapy students
  Interventions: Other: Clinical simulation

INTERVENTIONS:
Other: Clinical simulation — Carrying out a total of 9 clinical simulation in three days, one day a week, where the student resolves a situation by taking on the role of a physiotherapist with a simulated patient.

SUMMARY:
Clinical simulation has gained great importance in recent times in health sciences. Since it is a pedagogical strategy that is being used more and more in health degrees and is very useful for the acquisition of both technical and non-technical skills.

However, if we focus on physiotherapy, the use of clinical simulation is a very new field and therefore requires great research. The investigators still do not have the consistency or experience as in other health branches such as medicine or nursing, in which they have been using simulators for years for the learning of all their students.

For all this, and for the situation of need generated in recent years, in which internships in hospitals and clinical centers were completely abolished, the need for our research is justified, which will allow the acquisition of non-technical skills among novice students. in physiotherapy, without the need for contact with real patients.

ELIGIBILITY:
Inclusion Criteria:

* Second year students of the Physiotherapy Degree
* They do not have clinical experience with real patients.

Exclusion Criteria:

* Not wanting to sign to participate in the study.
* Not signing the informed consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 113 (Actual)
Dates: Start 2024-02-26 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Ottawa Scale | 1 week, 2, week, 3 week
  Modified Ottawa Scale for the acquisition of non-technical skills, validated in Spanish (https://doi.org/10.1016/j.redar.2021.02.009).
  Each of the items evaluated must be classified from 'strongly disagree', whose value is zero, to 'strongly agree', whose value is 7.
  The scale will be passed after each of the 9 simulations, which will be carried out 3 on the same day, for three weeks.

CONTACTS AND LOCATIONS:
Overall Officials: David Hernández-Guillén, Study Director — University of Valencia
Locations (1):
- David Hernández-Guillén, Valencia, Spain